CLINICAL TRIAL: NCT05845346
Title: Efficacy of Two Physiotherapy Intervention Methods Applied in Subjects in the Social-healthcare Setting With Nonspecific Neck Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Mª Ángeles Cardero Durán, Principal Investigator, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38/2014
Record Dates: First submitted 2023-02-23; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-02

CONDITIONS: Neck Pain
Keywords: inespecif pain; physicaltherapy
MeSH Terms: conditions — Neck Pain | interventions — Massage; Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group TENS (Experimental): Experimental group 1 will undergo a physiotherapy treatment based on TENS-type analgesic currents and application of massage therapy for neck pain.
  Interventions: Other: Electrotherapy-Transcutaneous Electrical Stimulation (TENS); Other: Massage therapy; Other: Ischaemic Compression Technique
- Group STRECHING (Experimental): Experimental group 2 will undergo a physiotherapy treatment based on stretching and the application of massage therapy therapy for neck pain.
  Interventions: Other: Massage therapy; Other: Stretching exercises; Other: Ischaemic Compression Technique
- Control Group (No Intervention): The control group will not undergo any physiotherapy treatment therapy for neck pain.

INTERVENTIONS:
Other: Electrotherapy-Transcutaneous Electrical Stimulation (TENS) — Ten electrotherapy sessions lasting 30 minutes were carried out. Analgesic currents of the TENS type, placed in the cervical region.
  Arms: Group TENS
Other: Massage therapy — Ten massage therapy sessions lasting 20 minutes each were carried out. Techniques such as superficial rubbing, deep rubbing, kneading and gliding pressure were performed on the cervical region.
  Arms: Group STRECHING; Group TENS
Other: Stretching exercises — Ten stretching exercise sessions.The stretching exercise modality performed consisted of passive static stretching with a sequence of 30s-10s-30s-10s.
  Arms: Group STRECHING
Other: Ischaemic Compression Technique — Ten Ischaemic Compression Technique sessions. The execution of the technique is described as follows: after locating a painful point (trigger point), pressure is applied until pain is generated, then a position is sought where the pain disappears, the position of maximum comfort, which is maintained for 90 seconds (sec), after which time the patient is returned to the starting position in a passive manner.
  Arms: Group STRECHING; Group TENS

SUMMARY:
The overall objective of this study is to compare the effectiveness of two physiotherapy treatments, one based on the application of massage most current analgesic TENS compared to a second massage treatment based on more specific stretching techniques in subject in th social-health care setting with non-specific neck pain.

DETAILED DESCRIPTION:
The subjects included in the sample will be evaluated according to the above-mentioned parameters by researchers trained and assigned for this purpose.

The data collection of the different variables will be carried out before and after the completion of the programs designed for the study. The programs designed for the experimental groups have a duration of 10 sessions, twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 18-60 years.
* Cervical pain of non-specific origin or Cervicalgia type I and II according to the Quebec - Task Force on Spinal Disorders.
* Be willing to participate in the study and sign the informed consent form.
* Have at least one year of seniority in the company exercising the current professional activity within the team of socio-health personnel.

Exclusion Criteria:

* Cervicalgia with neurological involvement or caused by pathologies such as: inflammatory disease, neurological disease, rheumatic disease, severe osteoporosis, fracture, dislocation, vertebro-basilar insufficiency, neoplasia or infection.
* Spine surgery.
* Present metallic implants at the spinal column level.
* Have received physiotherapy or alternative treatment in the last 6 months before starting the study.
* To present any type of inconvenience to the application of electrotherapy (score ≥45 points in EAPP).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain | 5 weeks
  A visual analog scale (VAS). The scale is represented by a 10 centimeter line on whose extremes have two adjectives, absence of pain and pain unbearable.
Changes in Range of Motion | 5 weeks
  Measurement of joint amplitude with goniometry. The ROM exploration was performed with the subjects in sitting in order to stabilize the pelvis and the thoracic-lumbar spine. From this position, the degrees of maximum position reached by the subjects in each of the 6 movements of space.
  Unit of measurement in degrees of articulation
Changes in Disability | 5 weeks
  Neck Disability Index through which will give us the degree of disability neck pain.The NDI consists of 10 sections, 4 of them are related to subjective symptoms (pain intensity, headache, head, ability to concentrate and quality of sleep) and the other 6 are related to ABVD (personal care, ability to lift weights, reading, work, driving, leisure activities and free time). Each of the sections presents 6 possible answers, scoring these from 0 to 5 according to the progression of functional disability.
General Health | 5 weeks
  The SF-12 contains 12 questions distributed in each of the 8 dimensions. The higher the score, the better the state of health.
Changes Pressure Pain | 5 weeks
  Pressure Pain with Algometry. To assess the mechanosensitivity of the trigger points , the pain threshold was measured at the pressure.
  Unit of measure Kg/cm2.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Espejo Antunez, Study Director — Universidad de Extremadura
Locations (1):
- María de los Ángeles Cardero Durán, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Covarrubias-Gomez A, Guevara-Lopez U, Lara-Solares A, Tamayo-Valenzuela AC, Salinas-Cruz J, Torres-Gonzalez R. [Clinical pattern of patients cared for at pain clinic by first time]. Rev Med Inst Mex Seguro Soc. 2008 Sep-Oct;46(5):467-72. Spanish. PMID 19241653
- [Background] Torres Cueco R. La columna cervical: síndromes clínicos y su tratamiento manipulativo. Ed panamericana. 2008; 233-234.
- [Background] Walker BF. The prevalence of low back pain: a systematic review of the literature from 1966 to 1998. J Spinal Disord. 2000 Jun;13(3):205-17. doi: 10.1097/00002517-200006000-00003. PMID 10872758
- [Background] Amer- Cuenca J.J. Programación y aplicación de la estimulación nerviosa eléctrica transcutanea (TENS): guía de práctica clínica basada en la evidencia. Fisioterapia 2010; 32(6):271-278.
- [Background] Fuentes JP, Armijo Olivo S, Magee DJ, Gross DP. Effectiveness of interferential current therapy in the management of musculoskeletal pain: a systematic review and meta-analysis. Phys Ther. 2010 Sep;90(9):1219-38. doi: 10.2522/ptj.20090335. Epub 2010 Jul 22. PMID 20651012
- [Background] Jonhoson MI, Tabasam G. A double blind placebo controlled investigation into the analgesic effects of inferential currents (IFC) and transcutaneous electrical nerve stimulation (TENS) on cold-induced pain in healthy subjects. Physiother Theory Pract 1999; 15: 217-33
- [Background] Calle Fuentes P, Muñoz- Cruzado y Barba M, Catalán Matamoros D, Fuentes Hervías M.T. Los efectos de los estiramientos musculares: ¿que sabemos realmente? Rev Iberoam Fisioter Kinesol 2006; 9(1):36-44.
- [Background] Meseguer-Henarejos, B, Medina-I-Mirapeix, F, Canovas-Gascón J.J, Esteban-Argente, I, Torres-Vaquero A.I, Alcántara F. Prevalencia, consecuencias y factores de riesgo de la cervicalgia. Fisioterapia. 2000; 22 (monográfico 2): 13-32

DOCUMENTS (1):
  • Informed Consent Form (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/46/NCT05845346/ICF_000.pdf